CLINICAL TRIAL: NCT05507190
Title: Self-management of Post COVID-19 Syndrome Using Wearable Biometric Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Diana C Sanchez-Ramirez, PhD, Assistant professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS25512(B2020:042
Record Dates: First submitted 2022-07-28; First posted 2022-08-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
Keywords: Long COVID-19; Persistent symptoms; Self-management
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm (Experimental): Self-management group. This pilot-study uses a one-group before-after design.
  Interventions: Other: Self-management of post COVID-19 respiratory outcomes

INTERVENTIONS:
Other: Self-management of post COVID-19 respiratory outcomes — Intervention: using the participants' initial assessment, personal characteristics, main complaints/needs and goals, the therapist will adjust the exercise plan and personalize the recommendations (e.g. maximum heart rate) as well as instruct the patients about safety precautions (how to pace themselves, when to seek professional or emergency care). Participants will be encouraged to wear the smart shirt as much as they want during the 6 weeks (29), but at a minimum of 1-hour a day (M-F) including while performing the recommended exercises (30-45 min/3 times a week). They should self-monitor their biometric values trying to reach/stay within the target values while wearing the shirt using Hexoskin app installed on an iPad provided by the research team or on the participants' personal device if preferred.

SUMMARY:
The main objective of this pilot study is to evaluate the impact of a self-management intervention using wearable biometric technology on post-COVID-19 syndrome. In addition, this pilot-study will provide information regarding validity, feasibility, patient compliance and satisfaction, valuable for the design of a future large-scale study.

DETAILED DESCRIPTION:
This pilot-study uses a one-group before-after design. Subjects: a convenience sample of 20 adults 18 years and older in the Winnipeg Health Region with a post-COVID-19 infection (≥ 3 months since acute infection) complaining of mild to severe persistent respiratory symptoms. Intervention: using the participants' initial assessment, personal characteristics, main complaints/needs and goals, the therapist will adjust the exercise plan and personalize the recommendations (e.g. maximum heart rate) as well as instruct the patients about safety precautions (how to pace themselves, when to seek professional or emergency care). Participants will be encouraged to wear the smart shirt as much as they want during the 6 weeks (29), but at a minimum of 1-hour a day (M-F) including while performing the recommended exercises (30-45 min/3 times a week). They should self-monitor their biometric values trying to reach/stay within the target values while wearing the shirt using Hexoskin app installed on an iPad provided by the research team or on the participants' personal device if preferred. Patients will also complete an online survey reporting symptoms intensity and activities completed, 3 times a week (over 6 weeks). Participants would be able to contact the research assistant overseeing the intervention at any time of the study if they have questions or concerns (text message or email). Otherwise, they will receive a follow-up phone call every week or if a significant change in their biometrical data is identified.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID-19 ≥ 3 months after infection.
* Mild to severe persistent respiratory symptoms
* Access to a home internet

Exclusion Criteria:

* History of neurological disease or mental illness
* Inability to ambulate independently without supervision
* Inability to complete basic tasks on a smart phone or tablet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in lung capacity | 6 weeks
  It will be assessed using a SpiroBank Smart F/V multi parameter spirometer (MIR) at pre-post intervention and once a week in between to monitor changes. This portable spirometer, which is MDSAP approved and complaint with ATS/ERS guidelines, connects automatically via Bluetooth to an iOS & Android compatible App (MIR Spirobank). It provides real time feedback through messages and animation on smartphone, to improve personal compliance during the test. The app can generate test results PDF printout with information regarding 19 parameters of lung capacity.
Change in dyspnea | 6 weeks
  Modified Borg Scale (0 "best" to 10 "worse dyspnea") will be used to assess dyspnea.
Change in fatigue | 6 weeks
  Fatigue severity scale (0 -7 "more fatigue") will be used to measure the severity of fatigue.
Chronic fatigue syndrome | 6 weeks
  DePaul Symptoms Questionnaire short form (DSQ-SF) (0 "not present" - 4 "very severe")
Health-related quality of life | 6 weeks
  EuroQol five-dimensional questionnaire (0 "worse health" to 100 "best health")
Postural orthostatic hypotension | 6 weeks
  Orthostatic Stress Test (Postural transitions)
Exercise capacity | 6 weeks
  The 6-min walk test (6 MWT) and the one-minute sit-to-stand test

SECONDARY OUTCOMES:
Symptoms change | 6 weeks
  Participants will be ask to rate their symptoms from 0-10 using an online form (base on the baseline symptoms)
Patient satisfaction with the study | 6 week
  Participants will complete a short summary with questions regarding their satisfaction with the study

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Centre, Winnipeg, Manitoba, Canada